CLINICAL TRIAL: NCT06874738
Title: A Real-world Clinical Study on the Treatment of Menopausal Syndrome With Liuwei Dihuang Pills
Status: Not yet recruiting | Type: Observational
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Lanxi Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Lianxin Wang, Principal Investigator, China Academy of Chinese Medical Sciences
Other Study IDs: Liuwei Dihuang Pills
Record Dates: First submitted 2025-02-14; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Menopausal Syndrome
Keywords: Liuwei Dihuang Pills; The real world; Efficacy; Clinical study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood,Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liuwei Dihuang Pills: The intervention in this cohort consisted of the Six-flavoured Dihuang Pill and the rest of the conventional treatment.
  Interventions: Drug: Liuwei Dihuang pills

INTERVENTIONS:
Drug: Liuwei Dihuang pills — Conventional treatment （Hormones, selective 5-hydroxytryptamine reuptake inhibitors, etc.）+ Liu Wei Di Huang Pills

SUMMARY:
To evaluate the clinical efficacy of the real-world Liuwei Dihuang pills for the treatment of female menopausal syndromes, and to provide a basis for effective, safe and rational clinical use of the drug.

DETAILED DESCRIPTION:
In this study, the patients were divided into exposed and non-exposed groups based on whether or not they were taking Liuwei Dihuang Pills.

The patients in the non-exposed group were treated routinely, and the patients in the exposed group were treated routinely + Liuwei Dihuang Pills. The patients in the exposed group were required to take the medication according to the dosage instructions for at least 4 consecutive weeks. Combined use of drugs is allowed without interfering with the treatment plan, and the use of drugs and combined use of drugs should be recorded truthfully, including the dose, duration, frequency, and so on. The type of drugs used in combination and the corresponding daily dose, daily frequency and duration of treatment. During the course of treatment, patients in both groups were required to receive follow-up assessment once every 4 weeks. Termination of the study included death, loss of patients, or achievement of study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45-55 years old
2. Patients with menopausal syndrome using Liuwei Dihuang Pills
3. Kidney Yin Deficiency Syndrome

Exclusion Criteria:

1. Individuals allergic to any components of the drug or excipients;
2. Individuals with other endocrine diseases;
3. Individuals with organic lesions of the reproductive system;
4. Individuals who have undergone bilateral oophorectomy, hysterectomy, or have ovarian dysfunction;
5. Individuals with endometrial hyperplasia or unexplained vaginal bleeding;
6. Individuals with malignant tumors, hematologic, or immune system diseases;
7. Individuals with severe cardiovascular, cerebrovascular, liver, or kidney diseases (e.g., serum transaminase levels more than 1.5 times the upper limit of normal, serum creatinine above the upper limit of normal);
8. Individuals with psychiatric disorders or dependence on alcohol or drugs;
9. Individuals with mental illness or communication barriers;
10. Individuals with other conditions that, in the investigator's judgment, may reduce the likelihood of enrollment or complicate the study process are not suitable for participation in this clinical research.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Menopausal syndrome refers to a series of physical and psychosomatic symptoms caused by the gradual decline of ovarian function and fluctuating or decreasing levels of sex hormones before and after menopause in women.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Menopausal Symptoms | 4 weeks
  The Kupperman Rating Scale is a global tool for assessing menopausal symptoms. It has 13 items covering common perimenopausal symptoms like hot flashes, sweating, paresthesia, insomnia, irritability, depression, dizziness, fatigue, arthralgia, headache, palpitations, formication, urinary infections, and sexual status. Each item is weighted and summed for a total score of 0-63. A lower score means more severe perimenopausal symptoms.The modified Kupperman Rating Scale will be used to assess menopausal symptoms. Participants will complete the questionnaire before, after treatment, and during follow-up. Researchers will calculate the total score.
Change of Hormone Levels | 4 weeks
  Sex hormone levels are key for evaluating the endocrine status of menopausal women. In patients with menopausal syndrome, sex hormone levels show elevated Follicle-Stimulating Hormone and Luteinizing Hormone, and reduced Estradiol. High Follicle-Stimulating Hormone points to ovarian dysfunction. Changes in the Luteinizing Hormone/Follicle-Stimulating Hormone ratio may be linked to polycystic ovary syndrome, and decreased Estradiol is associated with ovarian failure.

SECONDARY OUTCOMES:
Change of Quality in life | 4 weeks
  The Menopause-Specific Quality of Life Questionnaire assesses menopausal women's quality of life, covering four dimensions: vasomotor symptoms, psychosocial state, physical state, and sexual life, with 29 items in total. Each item is scored from 0 to 6, where 0 means no distress and 6 means extreme distress. The average score of items in each dimension is calculated. A higher score indicates lower quality of life in that dimension.
Change of TCM Syndrome Scores | 4 weeks
  The TCM syndrome score sheet, designed as per TCM theory, assesses menopausal patients' TCM syndromes, covering symptoms and signs inTCM, etc.Changes in TCM syndrome scores for menopausal syndrome reflect improvement or worsening. The scale uses a semi - quantitative grading method, assigning scores of 0, 1, 2, or 3 to represent the severity of symptoms in menopausal syndrome patients. The scores are added up to form the total syndrome score, with a minimum of 0 and a maximum of 42. A higher score means a more serious condition.

CONTACTS AND LOCATIONS:
Overall Officials: Lianxin Wang, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT06874738/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT06874738/ICF_001.pdf